CLINICAL TRIAL: NCT07093515
Title: A Cohort Study of Biomarkers, Risk Assessment, Imaging, and Neurodegeneration in Patients With Cerebral Small Vessel Disease
Brief Title: Biomarkers, Risk Assessment, Imaging, and Neurodegeneration in Cerebral Small Vessel Disease (BRAIN-CSVD)
Acronym: BRAIN-CSVD
Status: Not yet recruiting | Type: Observational
Sponsor: Zhejiang Hospital (Other)
Responsible Party: Principal Investigator, Junjun Wang, Senior Research Scientist, Zhejiang Hospital
Other Study IDs: BRAIN-CSVD
Record Dates: First submitted 2025-07-21; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Small Vessel Disease
MeSH Terms: conditions — Cerebral Small Vessel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with cerebral small vessel disease: Patients with at least one following imaging finding: white matter hyperintensities (Fazekas >or=1), lacune, cerebral microbleeds, recent small subcortical infarcts, or enlarged perivascular spaces (Grade 2 or more).
  Interventions: Other: No intervention
- Patients without cerebral small vessel disease: Patients without any following imaging finding: white matter hyperintensities (Fazekas >or=1), lacune, cerebral microbleeds, recent small subcortical infarcts, or enlarged perivascular spaces (Grade 2 or more).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The BRAIN-CSVD study is a single-center prospective cohort study focusing on cerebral small vessel disease (CSVD).Patients enrolled in this research will undergo assessments for vascular risk factors, cognitive and other neurological functions, neuroimaging, and biomarkers. The study aims to explore imaging and biomarker predictors of CSVD progression, and the pathophysiological mechanisms of CSVD.

DETAILED DESCRIPTION:
Cerebral small vessel disease (CSVD) is a common imaging finding in elderly population and can impair cognitive and other neurological functions. Radiologically, CSVD may manifest as white matter hyperintensities, lacunes, cerebral microbleeds, enlarged perivascular spaces and so on. Due to its complex imaging presentations and diverse neurological impacts, current preventive and therapeutic options for CSVD remain limited. This study involves collecting vascular risk factors, assessing global cognitive function, gait, and other neurological functions, performing multimodal MRI scans, and collecting blood samples from CSVD patients. The goal is to identify imaging markers and biomarkers that predict disease progression and to investigate the underlying pathophysiological mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old;
* Cerebral small vessel disease on MR imaging.

Exclusion Criteria:

* Cerebral infarction (except lacunar infarcts), cerebral hemorrhage, brain tumors, epilepsy, severe traumatic brain injury, or prior brain surgery;
* Secondary white matter hyperintensities due to inflammatory, toxic causes and so on;
* Contraindications to MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospital-based patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2030-12-30 (Estimated); Study Completion 2032-12-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive function | Follow-up assessments will be conducted at the 2nd year and 4th year
  Montreal Cognitive Assessment (MoCA) score, with a range of 0 to 30 points, where higher scores indicate better cognitive function.

SECONDARY OUTCOMES:
Stroke | Follow-up assessments will be conducted at the 2nd year and 4th year
  The rate of the patients with ischemic stroke or cerebral hemorrhagic stroke

IPD SHARING:
Plan to Share IPD: Undecided